CLINICAL TRIAL: NCT04396249
Title: Transcutaneous Vagus Nerve Stimulation for Cognitive Impairments in Community-Dwelling Elderly
Brief Title: tVNS for Cognitive Impairments in Community-Dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-64
Record Dates: First submitted 2020-05-10; First posted 2020-05-20 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Aging
Keywords: transcutaneous vagal nerve stimulation (tVNS); Aging; cognition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS group (Experimental): The active tVNS group will be stimulated with 10 sessions of active transcutaneous vagal nerve stimulation (tVNS)
  Interventions: Device: Active tVNS
- Sham tVNS group (Sham Comparator): The sham tVNS group will be stimulated with 10 sessions of sham transcutaneous vagal nerve stimulation (tVNS)
  Interventions: Device: Sham tVNS

INTERVENTIONS:
Device: Active tVNS — One electrode tip is used as their common terminal, and the other two electrode tips are respectively connected to the skin surfaces of the auricle and the external auditory meatus. Each subject will have 10 active tVNS sessions.The active tVNS group will be stimulated with a 2 mA current for 30 minutes.
  Arms: Active tVNS group
Device: Sham tVNS — Each subject will have 10 sham tVNS sessions.The sham tVNS group will be stimulated with a 2 mA current for 30 minutes. Except for the stimulation site, other parameters are the same as active group.
  Arms: Sham tVNS group

SUMMARY:
The goal of this study is to explore the effects of transcutaneous vagus nerve stimulation(tVNS) on improving cognition in community-dwelling elderly people. The study will recruit 120 subjects. Participants will undergo baseline cognitive assessment, EEG and eye tracking. Participants will be randomized to tVNS group and sham group. All subjects will repeat the baseline assessments after 1st session, 5th session，10th session and within 3 days after 10th session.

DETAILED DESCRIPTION:
Transcutaneous vagal nerve stimulation (tVNS) is a non-invasive neurostimulation technology.Recent studies have found that tVNS may involve in the regulation of cognition and improve the memory of the elderly.However, due to the limited number of studies, the effect of tVNS on improving cognitive function and stimulation parameters are currently unclear.

To investigate the effects of tVNS on improving cognition in community-dwelling elderly people, our study will recruit 120 subjects. Participants will undergo baseline cognitive assessment, EEG and eye tracking. Active vs. sham treatment will be randomly assigned in a 1:1 fashion in groups using computer generated lists. Subjects and evaluators will be blind to treatment. All subjects will repeat the baseline assessments after 1st session, 5th session，10th session and within 3 days after 10th session.

ELIGIBILITY:
Inclusion Criteria:

(1) 65≤age≤75 years old; (2) years of education ≥1 year; (3) normal daily life ability; (4) total score of The Chinese version of Mini-Mental State Examination (MMSE) : Non-illiterate group (not graduated from elementary school)> 14 points, elementary school group> 19 points, middle school and above group> 24 points).

Exclusion Criteria:

(1) People with obvious hearing, vision problems or communication difficulties; (2) People with obvious cognitive dysfunction (such as Alzheimer's disease); (3) People with serious medical diseases (such as heart disease, uremia, severe diarrhea) ; (4) In the stage of radiotherapy and chemotherapy; (5) People with serious neurological diseases (such as Parkinson's disease, infectious encephalopathy); (6) Patients with mental diseases (such as schizophrenia, depression, etc.); 7) Patients with substance abuse or alcohol dependence; (8) patients with implantable medical devices such as cardiac pacemakers; (9) patients with scars or inflammation on the ear skin.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
cognition | up to 2 weeks(end of the intervention)
  Identifying cognitive affected domains by using Cambridge Neuropsychological Test Automated Battery (CANTAB) (Memory:PAL、DMS、PRM; Executive Function : RTI、MOT)

SECONDARY OUTCOMES:
cognition | within 1 day after 1st session and 5th session and 1-week follow-up
  Identifying cognitive affected domains by using Cambridge Neuropsychological Test
PHQ-9 | up to 2 weeks(end of the intervention),1-week follow-up
  Patient Health Questionnaire-9 items，values:0-27, higher score indicates more severe depression symptoms
GAD-7 | up to 2 weeks(end of the intervention),1-week follow-up
  Generalized Anxiety Disorder-7，values:0-21, Higher score indicates more severe anxiety symptoms
Relative power for delta, theta, alpha, sensorimotor and lower beta frequency bands. | up to 2 weeks(end of the intervention)
  The power spectral density was calculated to extract the relative power for each frequency band and estimated as a log-ratio.
Antisaccade latency | up to 2 weeks(end of the intervention)
  We used an EyeLink Desktop 1000 eye-tracker to collect the information of eye movements.The latency of the saccade was measured from the onset of the saccade to the target onset.
Side-effects of tVNS | At each stimulation session, up to 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No